CLINICAL TRIAL: NCT02147275
Title: Monitoring Cerebral Oxygen Saturation in Hypertensive Patients Undergoing Major Abdominal Surgery
Brief Title: Monitoring Hypertensive Patients's Cerebral Oxygen Saturation
Acronym: MHPCOS
Status: Completed | Type: Observational
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Li Hongyi, Department of Anesthesiology, Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: TJH-AD-12888; 75888 (Other: Tongji hospital)
Record Dates: First submitted 2014-05-22; First posted 2014-05-26 (Estimated); Last update posted 2014-11-11 (Estimated); Status verified 2014-11

CONDITIONS: Surgical Complications From General Anesthesia; Hypertension; Cerebral Ischemia; Cerebral Anoxia
Keywords: hypertension; cerebral oxygen saturation; near-infrared spectroscopy; cognitive function
MeSH Terms: conditions — Hypertension; Brain Ischemia; Hypoxia, Brain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- hypertension disease: patients have hypertension disease, whether well-controlled or uncontrolled, more than 3 year

SUMMARY:
The purpose of this study is to determine whether there is a significant decrease in cerebral oxygen saturation in hypertensive patients undergoing major abdominal surgery and their correlation with standard monitoring parameters.

ELIGIBILITY:
Inclusion Criteria:

* patients have hypertension more than 3 year,whether well-controlled or uncontrolled,
* scheduled for major abdominal surgery for at least 2 h
* under general anesthesia
* American Society of Anesthesiologists（ASA）physical status : II ~ III
* Age > 30

Exclusion Criteria:

* pre-existing cerebral pathology for example episodes of cerebral ischemia or stroke;
* ASA physical status >IV
* hepatic failure
* renal failure
* preoperative Mini-Mental State Examination (MMSE) score less than 24
* a history of cardiovascular surgery or craniotomy
* cardiac failure
* respiratory failure

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients scheduled for major abdominal surgery such as gastrectomy, colon resection ,liver resection and duodenocephalo-pancreasectomy
Sampling Method: Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2014-05; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
decreases in cerebral oxygen saturation (rSO2) during the surgery | every 5 minutes throughout the surgery

SECONDARY OUTCOMES:
Change from baseline in Mini-Mental State Exam (MMSE) perioperative period | Baseline, 4 day after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Peng Wang, MD PHD, Study Director — Vice Director
Locations (1):
- Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

REFERENCES:
- [Derived] Li H, Fu Q, Wu Z, Sun J, Manyande A, Yang H, Wang P. Cerebral oxygen desaturation occurs frequently in patients with hypertension undergoing major abdominal surgery. J Clin Monit Comput. 2018 Apr;32(2):285-293. doi: 10.1007/s10877-017-0024-0. Epub 2017 May 9. PMID 28488169